CLINICAL TRIAL: NCT04438174
Title: A Phase I/II Clinical Trial To Determine Safety And Feasibility Of Using An Acellular Amniotic Fluid Application To Expedite Healing In Chronic Wounds
Brief Title: Processed Amniotic Fluid (pAF) for the Treatment of Chronic Wounds
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enrollment was halted prematurely after enrolling one participant due to difficulty finding eligible participants.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Giavonni Lewis, MD, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 128708
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: Wounds and Injuries
Keywords: chronic wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Wound digital images will be assessed and evaluated by two University Staff members blinded to both the control and treatment group (one primary and one secondary).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Amniotic Fluid Injection (Experimental): Processed Amniotic Fluid. Dose is 1ml/5cm2; Route: injected directly into wound; Limited to two injections. The wound will then be dressed according to standard of care.
  Interventions: Drug: Processed Amniotic Fluid
- Standard of Care Wound Treatment Regimen (Active Comparator): Primary dressings are variable and based on the moisture content and microorganism load. In general, wounds respond differently to various topical treatments. Through our clinical practice, we have found that wounds plateau with the same topical for greater than 4 weeks, hence changing antimicrobial topical helps to manage the bacterial overgrowth. We will start with our application of our slurry, a 1:1:1 ratio of Nystatin ointment, Mupirocin Ointment, and Bacitracin Ointment. This slurry will be applied directly to the cleansed wound, followed by silver gauze/foam product to all wounds. Types of silver product- site and comfort predict use of Restore, Mepilex-AG, or Mepitel-AG. If allergies to the above slurry occurs, we will use medical honey with or without bacitracin. If ointment related rash present with transition to silver product only or silver product plus medical honey.
  Interventions: Other: Standard of Care Wound Treatment Regimen

INTERVENTIONS:
Drug: Processed Amniotic Fluid — Injection of 1 ml of processed amniotic fluid per 5 cm2 of wound area
  Other Names: Processed Amniotic Fluids (pAF); Human Amniotic Fluids (hAF)
  Arms: Amniotic Fluid Injection
Other: Standard of Care Wound Treatment Regimen — ointment-based dressing and non-ointment-based dressings
  Arms: Standard of Care Wound Treatment Regimen

SUMMARY:
A prospective randomized controlled study to determine the safety and feasibility of using processed amniotic fluid (pAF) to expedite healing in chronic wounds.

DETAILED DESCRIPTION:
The goal of our study is to assess, in an outpatient setting, the safety and the time to wound closure in chronic wounds treated with processed amniotic fluid (pAF). We will include patients with lower extremity full thickness wounds that are greater than 3 months old and less than 12 months old. The wound size must be greater than 5cm2 and less than 75 cm2. We will exclude anyone that requires skin grafting, or wounds with sinus tracts. Our primary objective is to determine the safety and feasibility of using pAF to treat patients with chronic wounds. The secondary objective is to determine the efficacy of pAF compared to standard of care in reducing wound area.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18-85 years old.
2. Patients with chronic lower extremity wounds (including thermal) that are greater than 3 months, but less than 12 months old.
3. Patients with full thickness wounds.
4. Patients with at least one wound that is ≥5 cm2 and<75 cm2 in size.
5. Patient who is able to complete required site study visits and procedures in good faith

Exclusion Criteria:

1. Patients admitted to the hospital at the time of enrollment.
2. Patients who are pregnant, nursing or plan to become pregnant while participating in the study. If of child-bearing potential, unwillingness to use effective birth control while participating in the study.
3. Suspicion of or diagnosis of osteomyelitis underlying the wound.
4. Patients who have received an investigational agent or intervention within the prior 30 days or plan to use within the study period.
5. Patient with sinus tracts, enterocutaneous fistulas or other epithelialized tracts.
6. Patients who require skin grafting.
7. Patients diagnosed with a highly disruptive, non-controlled mental health disorder (e.g.., bipolar, or schizophrenia.
8. Patients with a history of prior drug abuse.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-08 (Actual); Primary Completion 2023-03 (Actual); Study Completion 2023-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giavonni Lewis, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Burn Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amniotic Fluid Injection | Standard of Care Wound Treatment Regimen
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrollment was halted prematurely after enrolling one subject.
Groups:
- Total: Total of all reporting groups
Arm/Group | Amniotic Fluid Injection | Standard of Care Wound Treatment Regimen | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants] — Age at randomization
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety - Adverse Events Including Serious Adverse Events
Description: Safety and tolerability will be evaluated by the PI from the results of reported signs and symptoms and scheduled physical examinations. The primary endpoint is whether the patient experienced any post-randomization, study-related serious adverse event (SAEs) while on study (collections of new AEs begins at visit two and ends at visit five which is approximately, 7 months after enrollment). An SAE is considered study-related if the medical monitor concludes the SAE is either possibly related or probably related to study participation. Although unresolved SAE's were to be monitored for 1 year or until resolution, no SAEs were unresolved at the time of study completion (approximately, 7 months after enrollment).
Time Frame: Approximately 7 months after enrollment
Population: Enrollment was halted prematurely after enrolling one participant due to difficulty finding eligible participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Amniotic Fluid Injection | Standard of Care Wound Treatment Regimen
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

2. Secondary Outcome: Feasibility - Reduction in Wound Size - Secondary Outcome Per Secondary Assessor
Description: The percent reduction in wound area at Visit 5 (final visit) relative to the size at randomization visit (visit 2). Wound surface area will be calculated and maximal wound depth will also be measured using ImageJ overlay software technology. Two assessors examined the wound surface area at each visit using ImageJ. This is the outcome as reported by the secondary assessor. A negative value indicates an increase in wound size; a positive value indicates a decrease in wound size.
Time Frame: Visit 2 (approximately 6 weeks after enrollment) and Visit 5 (approximately 7 months after enrollment)
Population: Enrollment was halted prematurely after enrolling one participant due to difficulty finding eligible participants.
Measure: Mean (Full Range); unit: percent reduction in wound area
Arm/Group | Amniotic Fluid Injection | Standard of Care Wound Treatment Regimen
Number analyzed (Participants) | 1 | 0
percent reduction in wound area | 91.4 [91.4 to 91.4] |

3. Secondary Outcome: Feasibility - Reduction in Wound Size - Secondary Outcome Per Primary Assessor
Description: The percent reduction in wound area at Visit 5 (final visit) relative to the size at randomization visit (visit 2). Wound surface area will be calculated and maximal wound depth will also be measured using ImageJ overlay software technology. Two assessors examined the wound surface area at each visit using ImageJ. This is the outcome as reported by the primary assessor. A negative value indicates an increase in wound size; a positive value indicates a decrease in wound size.
Time Frame: Visit 2 (approximately six weeks after enrollment) and Visit 5 (approximately 7 months after enrollment)
Population: Enrollment was halted prematurely after enrolling one participant due to difficulty finding eligible participants.
Measure: Mean (Full Range); unit: percent reduction in wound area
Arm/Group | Amniotic Fluid Injection | Standard of Care Wound Treatment Regimen
Number analyzed (Participants) | 1 | 0
percent reduction in wound area | -33.7 [-33.7 to -33.7] |

ADVERSE EVENTS:
Time Frame: For purposes of this study, events that occur following participant consent through visit 5 (approximately 7 months after enrollment) will be reported as adverse events.
Description: Adverse events were on the schedule of activities for collection at visits 2 through 5 (approximately 7 months after enrollment). Subjects were to receive a follow-up phone call within 24 hours AND 5-7 days after visit 2 and 3 to identify any adverse events that occur in relation to study participation and record additional medications that were taken.
Arm/Group | Amniotic Fluid Injection | Standard of Care Wound Treatment Regimen
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amniotic Fluid Injection (N=1) | Standard of Care Wound Treatment Regimen (N=0)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amniotic Fluid Injection (N=1) | Standard of Care Wound Treatment Regimen (N=0)
Wound drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Gram stain positive (Investigations) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ulcer (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment was halted prematurely after successful enrollment of one participant due to limited eligible participants. A single participant was enrolled in the treatment arm, hence we are unable to measure the safety and effectiveness of the intervention compared to standard care. We noted variation in wound size assessment for our single participant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT04438174/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT04438174/SAP_001.pdf
  • Informed Consent Form (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT04438174/ICF_003.pdf